CLINICAL TRIAL: NCT04008537
Title: A Pilot Study of Daily Imaging, Target Identification, and Simulated Computed Tomography-Based Stereotactic Adaptive Radiotherapy Workflow in a Novel Ring Gantry Radiotherapy Device
Brief Title: Daily Imaging, Target Identification, and Simulated Computed Tomography-Based Stereotactic Adaptive Radiotherapy Workflow in a Novel Ring Gantry Radiotherapy Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201908024
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Cancer of Pancreas; Cancer of Pelvis; Cancer of Abdomen; Cancer of Thorax
MeSH Terms: conditions — Pancreatic Neoplasms; Pelvic Neoplasms | interventions — Particle Accelerators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Halcyon kV CBCT imaging (Experimental): -Each patient will undergo five Halcyon kV CBCT imaging sessions that will then be utilized to simulate the CBCT-guided online ART workflow. Halcyon imaging will be scheduled as per the patient's schedule and availability, with intent but not mandate for imaging on the same days as clinical treatments, preceding clinical treatment. Multiple images may be acquired in one session but no more than 6 Halcyon kV CBCT images will be acquired per day. No more than 6 additional Halcyon kV CBCT images will be acquired in one imaging session and no more than 10 total additional Halcyon kV CBCT images for the duration of the study
  Interventions: Device: Ring gantry kV-CBCT combined with linear accelerator

INTERVENTIONS:
Device: Ring gantry kV-CBCT combined with linear accelerator — Each imaging session will be less than one hour, and is expected to take no more than 15 minutes.
  Other Names: Halcyon

SUMMARY:
The investigators propose here to evaluate the feasibility of a novel cone-beam CT (CBCT)-guided online adaptive radiotherapy (ART) workflow on the Halcyon device.

ELIGIBILITY:
Inclusion Criteria:

* At least one disease site deemed to be suitable for simulated treatment with online adaptive radiotherapy per radiation oncology evaluation.
* Scheduled to receive radiation therapy to the thorax (n = 8), pancreas (n = 8), non-pancreas abdomen (n = 8), or pelvis (n = 8).
* At least 18 years of age
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry. If pregnancy test is not clinically indicated as determined by treating physician or protocol PI, documentation of this exception is sufficient in lieu of a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the device as measured by successful completion of the full CBCT-guided online ART workflow, from volumetric imaging through phantom delivery in at least 90% of attempted fractions | Completion of ART workflow in all enrolled participants (estimated to be 30 months)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Henke, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu